CLINICAL TRIAL: NCT04491812
Title: Role of Triceps Kinesiology Taping on Elbow Flexion Tightness in Extended Erb's Palsy Infants
Brief Title: Triceps Taping on Elbow Flexion Tightness in Extended Erb's Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Radwa Said, Principal Investigator, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P.T.REC/012/001922
Record Dates: First submitted 2020-07-16; First posted 2020-07-29 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Deformity Flexion
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Group A: physical therapy program Group B: physical therapy program inaddition to kinesiotaping
Who Masked: Participant
Masking Description: single blind masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping (Experimental): kinesiotaping of the triceps muscle applied to the study group alongside the physical therapy program
  Interventions: Other: Kinesio Tape
- physical therapy program (Placebo Comparator): the control group recieved only the physical therapy program
  Interventions: Other: Physical therapy program

INTERVENTIONS:
Other: Kinesio Tape — Elastic Kinesiology Tape
  Arms: Kinesiotaping
Other: Physical therapy program — designed physical therapy program
  Arms: physical therapy program

SUMMARY:
To determine the role of using Kinesiology tape on the prevention of elbow flexion tightness in infants with extended Erb's palsy.

DETAILED DESCRIPTION:
PURPOSE:

To determine the role of using Kinesiology tape on the prevention of elbow flexion tightness in infants with extended Erb's palsy.

BACKGROUND:

BACKGROUND Neglecting or even delay in Brachial plexus birth palsy management, may result in substantial and chronic impairment. Physiotherapy, microsurgical nerve reconstruction, secondary joint corrections, and muscle transpositions are employed to help the child maximize function in the affected upper extremity. Kinesiology taping can have an effect on muscle performance and support joint by improving proprioception, normalizing muscle tone, correct the inappropriate positions and stimulate skin receptors. The possible effect of kinesiotaping on muscle strength has been investigated by numerous researchers that have theorized that kinesiotaping facilitates an immediate increase in muscle strength by generating a concentric pull on the fascia.

HYPOTHESES:

There will be no role of Kinesiology tape on the prevention of elbow flexion tightness in infants with extended Erb's palsy.

RESEARCH QUESTION:

Is there a role of using Kinesiology tape in preventing elbow flexion tightness in infants with extended Erb's palsy?

ELIGIBILITY:
Inclusion Criteria:

* 3-6 months of age
* had unilateral extended BPBP involving cervical 5, 6, and 7 roots lesion
* based on an EMG referral by a physiatrist
* had positive grasp reflex on both sides
* had asymmetrical Moro reflex on the affected side.

Exclusion Criteria:

- surgical interferences arm fracture or dislocations hypersensitivity to latex and adhesive tapes

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-09-10 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Elbow extension ROM | 3 months
  The range of motion of the extension of the elbow will be measured by smartphone goniometer "G-Pro" and recorded in "degrees"

SECONDARY OUTCOMES:
muscle strength | 3 months
  elbow flexors and extensors muscle strength will be measured using the "Toronto Active Movement Scale" and recorded by number scale from 0-7; 0 meaning no contraction while 7 mean normal power

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty pf physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-05-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT04491812/Prot_ICF_000.pdf